CLINICAL TRIAL: NCT00730652
Title: A Phase I, Open-Label, Multicenter, Dose-escalation, Multidose Study of MDX-1411 Administered Every 7 Days in Subjects With Relapsed/Refractory Chronic Lymphocytic Leukemia or Mantle Cell Lymphoma
Brief Title: Study of MDX-1411 in Patients With Relapsed/Refractory Chronic Lymphocytic Leukemia or Mantle Cell Lymphoma
Acronym: MDX1411-02
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MDX1411-02
Record Dates: First submitted 2008-08-04; First posted 2008-08-08 (Estimated); Last update posted 2010-04-22 (Estimated); Status verified 2010-04

CONDITIONS: Chronic Lymphocytic Leukemia or Mantle Cell Lymphoma.
Keywords: Medarex Inc.
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Mantle-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MDX1411 (Experimental): An accelerated titration design (ATD) will be utilized and subjects will be assigned to a dose level in the order they enter the study.
  Interventions: Biological: MDX-1411

INTERVENTIONS:
Biological: MDX-1411 — Single dose of MDX-1411 (fully human monoclonal antibody) will be administered as an intravenous (i.v.) infusion every 7 days for up to a total of 5 doses.

SUMMARY:
To determine if MDX-1411 is safe for the treatment of chronic lymphocytic leukemia or mantle cell lymphoma.

DETAILED DESCRIPTION:
Dose-escalation, multidose study of MDX-1411, a fully human nonfucosylated monoclonal antibody (mAb) targeting the CD70 transmembrane cell-surface protein, which is highly expressed in B-cell malignancies such as CLL and MCL.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of relapsed/refractory MCL or hematologically/bone marrow confirmed relapsed/refractory CLL that is not amenable to cure by surgery or other means and has failed at least 1 prior systemic therapy;
* Subjects may have been treated with up to 6 prior systemic therapies for relapsed/refractory disease or have become intolerant to a systemic therapy
* For MCL, must have measurable disease
* At least 4 weeks since the last systemic therapy, including RT, for the treatment of MCL/CLL;
* At least 4 weeks since taking any corticosteroids prior to the first dose of MDX-1411
* ECOG Performance Status 0 to 2;
* No known positivity for human immunodeficiency virus (HIV) and no active infection with Hepatitis B or Hepatitis C;

Exclusion Criteria:

* History of severe hypersensitivity reactions to other monoclonal antibodies;
* Use of other investigational drugs within 30 days before study drug administration
* Prior treatment with any other anti-CD70 antibody;
* Active infection requiring i.v. systemic therapy within 4 weeks of receiving the first dose of MDX-1411;
* Evidence of bleeding diathesis or coagulopathy;
* Active autoimmune disease requiring immunosuppressive therapy;
* Known current drug or alcohol abuse;
* Underlying medical conditions that will make the administration of MDX-1411 hazardous

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2009-05; Primary Completion 2012-12 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
Safety Profile of MDX-1411 and determine the maximum tolerated dose (MTD) | Day 1-40

CONTACTS AND LOCATIONS:
Overall Officials: Medarex Medical Monitor, Study Director — Medarex